CLINICAL TRIAL: NCT05498246
Title: Bipolar Coagulation Versus Suture Renorrhaphy for Hemostasis of Tumour Bed in Laparoscopic Partial Nephrectomy: Prospective Randomized Comparative Study
Brief Title: Bipolar Coagulation Versus Suture Renorrhaphy in Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed Kadry Mostafa, Bipolar coagulation versus suture renorrhaphy for hemostasis of tumour bed in laparoscopic partial nephrectomy: prospective randomized comparative study, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lap in partial nephrectomy
Record Dates: First submitted 2022-08-03; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Nephrectomy

STUDY DESIGN:
Intervention Model Description: Patients were divided into two groups by close envelope method in this prospective study. group (A) included 30 cases in which we used bipolar coagulation for hemostasis ,group (B) included 30 cases in which we used suture renorrhaphy.
Who Masked: Participant
Masking Description: Patients were divided into two groups by close envelope method in this prospective study. group (A) included 30 cases in which we used bipolar coagulation for hemostasis ,group (B) included 30 cases in which we used suture renorrhaphy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (A) included 30 cases in which we used bipolar coagulation for hemostasis (Active Comparator): group (A) included 30 cases in which we used bipolar coagulation for hemostasis
  Interventions: Procedure: laparoscopic partial nephrectomy
- group (B) included 30 cases in which we used suture renorrhaphy (Active Comparator): group (B) included 30 cases in which we used suture renorrhaphy
  Interventions: Procedure: laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: laparoscopic partial nephrectomy — Operations were done under general anesthesia. Patients were positioned in modified lateral kidney position for trans-peritoneal procedures. Pneumoperitoneum using the Veress needle technique and trocar placement . Dissection to the renal hilum for good and sufficient exposure of the renal vessels. Good exposure of the tumor and marking the excision site with electro cautery. Clamping of renal vessels using laparoscopic Bulldog appliers. Excision of the renal mass using visual assessment to determine the suitable depth of normal parenchyma to be excised in order to achieve a negative surgical margin. Unclamping was done and re-assessment of the hemostasis to secure residual bleeding points. Approximation of the edges of renal parenchyma using suturing in both groups. The specimen was placed in an EndoCatch bag and removed through pfannenstiel incisionsurgical drain was placed in the paracolic gutter

SUMMARY:
To compare between bipolar coagulation of tumor bed in laparoscopic partial nephrectomy versus suture renorrhaphy

DETAILED DESCRIPTION:
Partial nephrectomy is the standard of care for T1 renal masses (local tumour) it preserves as much normal renal tissue as possible to avoid post-operative acute renal failure, chronic kidney disease and associated metabolic and cardiovascular morbidities . The main challenges that affect partial nephrectomy outcome is the need for renal ischemia to achieve good hemostasis, and the long-term oncological consequences associated with positive surgical margin. Laparoscopic partial nephrectomy has been widely used lately as it is associated with less blood loss, short hospital stay and early recovery in comparison to open partial nephrectomy . Hemostasis of the tumor bed after laparoscopic partial nephrectomy can be achieved by various techniques including Suture renorrhaphy which can be used whatever the bleeding area, the size of bleeding vessel, or the amount of bleeding. However, it consumes more ischemia time, involves functional parenchyma, and requires high laparoscopic skills . There for in our study we tried to find a way to improve the functional and oncological outcome of laparoscopic partial nephrectomy by comparing the bipolar coagulation versus conventional suture renorrhaphy in performing stable hemostasis of tumor bed

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of renal mass less than 7cm
* Renal mass in patients with chronic kidney disease

Exclusion Criteria:

* Patients with Central or hilar renal masses
* Renal masses close to pelvi-calyceal system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
To compare between bipolar coagulation of tumor bed in laparoscopic partial nephrectomy versus suture renorrhaphy | baseline frame
  patients were assessed preoperative by weight in kg and height in meters weight and height will be combined to report body mass index in kg/m^2 ,base line creatinine in mil gm ,baseline hemoglobin in gm,leterality ,CT to examine size in cm and RENAL score and asses patients intra operative by operative time in minutes ,ischemic time in minutes ,estimated blood loss in gm and hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: mostafa khalil, MD, Principal Investigator — Data analysis; Ali Abdelkarim, MD, Principal Investigator — data collections
Locations (1):
- Mohamed Kadry Mostafa, Banhā, Qalyubia Governorate, Egypt

REFERENCES:
- [Result] Msezane LP, Katz MH, Gofrit ON, Shalhav AL, Zorn KC. Hemostatic agents and instruments in laparoscopic renal surgery. J Endourol. 2008 Mar;22(3):403-8. doi: 10.1089/end.2007.9844. PMID 18355135
- [Result] Aron M, Gill IS. Minimally invasive nephron-sparing surgery (MINSS) for renal tumours part I: laparoscopic partial nephrectomy. Eur Urol. 2007 Feb;51(2):337-46; discussion 46-7. doi: 10.1016/j.eururo.2006.10.018. Epub 2006 Oct 20. PMID 17095144
- [Result] Zhang C, Xu Y, Zhang Z, Qiao B, Yang K, Liu R, Ma B. Laparoscopic simple enucleation and coagulation on tumor bed using argon beam coagulator for treating small renal cell carcinomas: an animal study followed by clinical application. Med Sci Monit. 2012 May;18(5):BR193-7. doi: 10.12659/msm.882729. PMID 22534702
- [Result] Harbin, A. C, Giusto, L, Lee, V. S., Nadhan, K., Mooney, J., & Eun, D. D. The Use of Argon Beam Coagulation During Robotic Partial Nephrectomy in an Animal Model. Videourology. (2015).
- [Result] Garcia-Segui A, Bercowsky E, Gascon-Mir M. [Simplified renorrhaphy using self-retaining barbed suture during laparoscopic partial nephrectomy]. Actas Urol Esp. 2012 Sep;36(8):497-502. doi: 10.1016/j.acuro.2012.04.001. Epub 2012 Jul 20. Spanish. PMID 22819349
- [Result] Campbell SC, Novick AC, Belldegrun A, Blute ML, Chow GK, Derweesh IH, Faraday MM, Kaouk JH, Leveillee RJ, Matin SF, Russo P, Uzzo RG; Practice Guidelines Committee of the American Urological Association. Guideline for management of the clinical T1 renal mass. J Urol. 2009 Oct;182(4):1271-9. doi: 10.1016/j.juro.2009.07.004. Epub 2009 Aug 14. No abstract available. PMID 19683266
- [Result] Kutikov A, Uzzo RG. The R.E.N.A.L. nephrometry score: a comprehensive standardized system for quantitating renal tumor size, location and depth. J Urol. 2009 Sep;182(3):844-53. doi: 10.1016/j.juro.2009.05.035. Epub 2009 Jul 17. PMID 19616235
- [Result] Moinzadeh A, Gill IS, Rubenstein M, Ukimura O, Aron M, Spaliviero M, Nahen K, Finelli A, Magi-Galluzzi C, Desai M, Kaouk J, Ulchaker JC. Potassium-titanyl-phosphate laser laparoscopic partial nephrectomy without hilar clamping in the survival calf model. J Urol. 2005 Sep;174(3):1110-4. doi: 10.1097/01.ju.0000168620.36893.6c. PMID 16094075
- [Result] Harmon WJ, Kavoussi LR, Bishoff JT. Laparoscopic nephron-sparing surgery for solid renal masses using the ultrasonic shears. Urology. 2000 Nov 1;56(5):754-9. doi: 10.1016/s0090-4295(00)00766-4. PMID 11068293
- [Result] Desai MM, Gill IS, Ramani AP, Spaliviero M, Rybicki L, Kaouk JH. The impact of warm ischaemia on renal function after laparoscopic partial nephrectomy. BJU Int. 2005 Feb;95(3):377-83. doi: 10.1111/j.1464-410X.2005.05304.x. PMID 15679798
- [Result] Zhao PT, Richstone L, Kavoussi LR. Laparoscopic partial nephrectomy. Int J Surg. 2016 Dec;36(Pt C):548-553. doi: 10.1016/j.ijsu.2016.04.028. Epub 2016 Apr 21. PMID 27109204
- [Result] Ota T, Komori H, Rii J, Ochi A, Suzuki K, Shiga N, Nishiyama H. Soft coagulation in partial nephrectomy without renorrhaphy: feasibility of a new technique and early outcomes. Int J Urol. 2014 Mar;21(3):244-7. doi: 10.1111/iju.12276. Epub 2013 Sep 18. PMID 24102735
- [Result] Kim DK, Kim LH, Raheem AA, Shin TY, Alabdulaali I, Yoon YE, Han WK, Rha KH. Comparison of Trifecta and Pentafecta Outcomes between T1a and T1b Renal Masses following Robot-Assisted Partial Nephrectomy (RAPN) with Minimum One Year Follow Up: Can RAPN for T1b Renal Masses Be Feasible? PLoS One. 2016 Mar 17;11(3):e0151738. doi: 10.1371/journal.pone.0151738. eCollection 2016. PMID 26987069
- [Result] Ramani AP, Desai MM, Steinberg AP, Ng CS, Abreu SC, Kaouk JH, Finelli A, Novick AC, Gill IS. Complications of laparoscopic partial nephrectomy in 200 cases. J Urol. 2005 Jan;173(1):42-7. doi: 10.1097/01.ju.0000147177.20458.73. PMID 15592022
- [Result] Takagi T, Kondo T, Omae K, Iizuka J, Kobayashi H, Yoshida K, Hashimoto Y, Tanabe K. Assessment of Surgical Outcomes of the Non-renorrhaphy Technique in Open Partial Nephrectomy for >/=T1b Renal Tumors. Urology. 2015 Sep;86(3):529-33. doi: 10.1016/j.urology.2015.05.018. Epub 2015 Jul 14. PMID 26187014
- [Result] Marszalek M, Chromecki T, Al-Ali BM, Meixl H, Madersbacher S, Jeschke K, Pummer K, Zigeuner R. Laparoscopic partial nephrectomy: a matched-pair comparison of the transperitoneal versus the retroperitoneal approach. Urology. 2011 Jan;77(1):109-13. doi: 10.1016/j.urology.2010.02.057. PMID 20970830
- [Result] Williams SB, Kacker R, Alemozaffar M, Francisco IS, Mechaber J, Wagner AA. Robotic partial nephrectomy versus laparoscopic partial nephrectomy: a single laparoscopic trained surgeon's experience in the development of a robotic partial nephrectomy program. World J Urol. 2013 Aug;31(4):793-8. doi: 10.1007/s00345-011-0648-5. Epub 2011 Jan 29. PMID 21274541